CLINICAL TRIAL: NCT06269640
Title: NHLBI SESAME (SEptal Scoring Along Midline Endocardium) Early Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Clinical trials terminated early due to trial feasibility
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001640; 001640-H
Record Dates: First submitted 2024-02-17; First posted 2024-02-21 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Cardiomyopathy; Left Ventricular Septal Hypertrophy; Mitral Valve Disease; Aortic Valve Stenosis
Keywords: transcatheter electrosurgery; transcatheter ventricular myotomy; Cardiac interventricular septal reduction
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure (Experimental): Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure that relies on intramyocardial guidewire navigation and transcatheter electrosurgery.
  Interventions: Device: Septal Scoring Along Midline Endocardium

INTERVENTIONS:
Device: Septal Scoring Along Midline Endocardium — Transcatheter ventricular myotomy called SEptal Scoring Along the Midline Endocardium (SESAME) that relies on intramyocardial guidewire navigation and transcatheter electrosurgery

SUMMARY:
Background:

Some people have a condition in which the wall (septum) that separates the two main pumping chambers of the heart is too thick. This thick septum causes a condition called "left ventricular outflow tract obstruction" (LVOTO), which reduces blood flow out of the heart. LVOTO can cause serious heart disease; symptoms may include shortness of breath, chest pain, heart failure, or death. Researchers want to find better ways to treat LVOTO.

Objective:

To test a new procedure where excess tissue is sliced away from the septum in people with LVOTO. This procedure is called "septal scoring along midline endocardium" (SESAME).

Eligibility:

Adults aged 21 years with LVOTO.

Design:

Participants will have baseline tests. They will have imaging scans and tests of their heart structure and function. They will take a walking test and answer questions about how their heart condition affects their life.

Participants will stay in the hospital 2 to 6 days for the SESAME procedure.

They will be completely or partially asleep for the procedure. A tube will be inserted into the mouth and down the throat to take pictures of the heart. Pictures may also be taken with a tube inserted inside the heart.

Next, tubes will be inserted into the groin and guided through the blood vessels up to the heart. Guidewires will be inserted into the heart. Doctors will watch the path the wires take with x-rays and ultrasound. When the wire is in the correct place, it will be electrified to slice excess tissue away from the septum.

Participants will have 3 follow-up visits within 1 year.

DETAILED DESCRIPTION:
Cardiac interventricular septal reduction therapies - to relieve left ventricular outflow tract obstruction from transcatheter valve replacement or hypertrophic cardiomyopathy - have inherent limitations including dependence on coronary anatomy, high pacemaker implantation rate, and surgical morbidity. We developed a novel transcatheter ventricular myotomy called SEptal Scoring Along the Midline Endocardium (SESAME) that relies on intramyocardial guidewire navigation and transcatheter electrosurgery. SESAME has been performed on a small number of patients using off label devices.

This study systematically characterizes the safety and early feasibility of SESAME at 2 enrolling site. SESAME is performed as septal reduction therapy in a heterogeneous group of subjects, including symptomatic hypertrophic cardiomyopathy and resting or provoked left ventricular outflow obstruction (LVOTO); and severe symptomatic mitral and/or aortic valve disease at high risk of standard heart surgical therapy and requiring later transcatheter heart valve implantation combined with manifest or potential LVOTO.

A key goal of this study is to attempt to capture generalizable knowledge from as many patients as possible, and to add a limited number of research procedures to characterize the safety and provisional effectiveness of SESAME. Absent realistic non-clinical models of HCM or LVH combined with aortomitral disease, we believe little more information can be gleaned without clinical investigation.

This protocol was revised to add a second enrolling medical center, and to focus inclusion criteria on research participants with hypertrophic cardiomyopathy (HCM). This protocol was further revised after the first subject died as a result of excessively-deep SESAME laceration. The required septal thickness for eligibility was increased from >=12mm to >=16mm.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults age >= 21 years
* Requires debulking of left ventricular septum for hypertrophic cardiomyopathy
* Septal diastolic thickness of obstructive hump on CT:

  * Total >=16 mm, and
  * Predicted residual septal thickness >= 8 mm, and
  * Predicted laceration depth >= 6 mm
* Severely symptomatic, any of

  * NYHA Class III or greater
  * Canadian Angina Class CCS III or greater
* Explicitly chooses investigational SESAME over conventional treatment approaches including (1) cardiac myosin inhibitor therapy, if eligible; (2) transcoronary alcohol septal ablation, if eligible; or (3) surgical left ventricular myotomy and/or myectomy, if eligible
* Concurrence of the multidisciplinary institutional heart team that the candidate is at high risk for surgical myectomy
* Concurrence of the study Central Clinical Eligibility Committee
* Willing to return for all scheduled follow-up activities, and eligible or able to undergo required protocol and testing

EXCLUSION CRITERIA:

* Does not consent to participate, or unable to consent to participate
* Requires antegrade SESAME access (because of mechanical aortic valve)
* Prior completed transcoronary alcohol septal ablation, or prior surgical myectomy
* Pregnant
* Hemodynamic instability or emergency procedure
* eGFR < 30 mL/min/1.73m^2
* Survival despite successful procedure expected < 12months

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
A peer-reviewed manuscript will constitute the clinical study report and shared data in Figshare after the manuscript is published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon acceptance of the peer-reviewed manuscript.
Access Criteria: unrestricted

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant That Experienced Technical Success With the SESAME (SEptal Scoring Along Midline Endocardium)
Description: The primary feasibility endpoint is Technical success with the SESAME (SEptal Scoring Along Midline Endocardium) technique.
  All of the following must be present:
  * Alive
  * Procedure success including
  * Successful myocardial entry, navigation, and snaring of guidewire traversal system; and
  * Successful laceration of septal myocardium
Time Frame: 1 minute following procedure discharge (Exit from the catheterization laboratory)
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Number of Inpatient Safety Events Related to SESAME (SEptal Scoring Along Midline Endocardium)
Description: Number of Inpatient Safety Events related to SESAME (SEptal Scoring Along Midline Endocardium)
  Safety is measured as freedom from all of the following:
  * All-cause mortality
  * All stroke (disabling and non-disabling)
  * Major cardiac structural complication requiring intervention (such as iatrogenic ventricular septal defect, iatrogenic aortic valve regurgitation, iatrogenic mitral regurgitation, or pericardial tamponade).
Time Frame: Up to 4 days
Measure: Number; unit: Number of Safety Events
Arm/Group | Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure
Number analyzed (Participants) | 1
Number of Safety Events | 2

3. Secondary Outcome: Number of Complete Heart Block Events
Description: Number of Complete heart block events requiring permanent pacemaker included in cardiac arrest
Time Frame: Up to 4 Days
Measure: Number; unit: Complete Heart Block Events
Arm/Group | Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure
Number analyzed (Participants) | 1
Complete Heart Block Events | 1

ADVERSE EVENTS:
Time Frame: Up to 4 days
Arm/Group | Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Undergoing SEptal Scoring Along Midline Endocardium (SESAME) Procedure (N=1)
Multipressor Vasoplegic Shock (General disorders) | 1 (1)
Ventricular Septal Defect (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may not independently publish, present, or disclose study results, in whole or in part, without permission of the Publications Committee.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT06269640/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT06269640/ICF_001.pdf